CLINICAL TRIAL: NCT05757206
Title: Cutaneous Phosphorylated Alpha-Synuclein for Detection of Prodromal Synucleinopathies
Brief Title: The Syn-Sleep Study
Status: Active, not recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 102
Record Dates: First submitted 2023-02-17; First posted 2023-03-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: REM Sleep Behavior Disorder (iRBD)
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Syn-One Test — Participating subjects will have three small skin punch biopsies.

SUMMARY:
In collaboration with approximately 8 centers that specialize in iRBD we will recruit a total of 80 individuals for the study. All subjects will be enrolled into a 2-year longitudinal study where skin biopsies will be performed at 3 sites on each patient at 12-month intervals (baseline, year 1, year 2). Plasma blood collection will be performed at 12-month intervals (baseline, year 1, year 2). Detailed quantified examination, cognitive evaluation, medical history, and questionnaires will be performed at each visit. Additional biomarker, imaging and clinical information (if available) will be obtained for the purpose of determining phenoconversion to clinically apparent synucleinopathy.

Subjects enrolled in the study will have baseline evaluations and follow up visits at 12 and 24 months to define any changes to clinical diagnosis (clinical phenoconversion). Skin biopsies will be repeated at the 12- and 24-month follow up visits to determine the rate of P-SYN accumulation over time and the rates of nerve fiber degeneration within punch skin biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-85
2. Subjects will have repeated episodes of sleep related vocalizations and/or complex motor behaviors
3. Sleep-related behaviors/disturbances must be documented by polysomnography to occur during REM sleep
4. Polysomnographic recording is consistent with REM sleep without atonia

Exclusion Criteria:

1. Subjects with MoCA < 19, Hoehn and Yahr score >/=1, contraindications to skin biopsy
2. Diagnosis of Parkinson's disease
3. Diagnosis of dementia of any type
4. Diagnosis of multiple system atrophy
5. REM sleep behaviors/disturbances secondary to another cause (e.g., narcolepsy, dementia, and Parkinson's disease)
6. Contra-indications to skin biopsy:

   1. Clinical evidence of severe vascular disease (history of ulceration, poor wound healing, and vascular claudication)
   2. History of allergic reaction to local anesthesia for skin biopsies
   3. Use of blood thinners (aspirin of Plavix alone is allowed)
   4. Significantly impaired wound healing or history of scarring or keloid formation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender at birth
Study Population: 80 subjects diagnosed with iRBD
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Advance the diagnostic utility of the Syn-One Test | 3 years
  Advance the diagnostic utility of the Syn-One Test™ by defining the metrics of P-SYN deposition and nerve fiber degeneration that predict phenoconversion in iRBD patients.
Enhance pathological reading through digital quantitative analysis of the Syn-One Test | 3 years
  Enhance pathological reading through digital quantitative analysis of the Syn-One Test™ using an AI-augmented detection system. Whole slide imaging with extraction of representative neural structures, target stain detection, segmentation, stain quantification and pattern recognition will be performed using deep learning algorithms. Results will be compared against pathologist readings and actual follow-up data to further refine model accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Levine, Principal Investigator — CND Life Sciences
Locations (8):
- United States (8):
  - MD First Research, Chandler, Arizona
  - Banner Health, Phoenix, Arizona
  - CND Life Sciences, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - University of Kentucky, Lexington, Kentucky
  - Mount Sinai, New York, New York
  - Texas Institute for Neurological Disorders, Sherman, Texas

IPD SHARING:
Plan to Share IPD: Undecided